CLINICAL TRIAL: NCT04886856
Title: Mindful Moms Randomized Control Trial Study
Brief Title: Mindful Moms Randomized Control Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM20021720; 1R01NR020220 (NIH)
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Depression
Keywords: pregnancy
MeSH Terms: conditions — Depression | interventions — Prenatal Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Moms (Experimental): Weekly "Mindful Moms" sessions
  Interventions: Behavioral: Mindful Moms
- Prenatal Education (Active Comparator): Weekly prenatal education sessions
  Interventions: Behavioral: Prenatal Education

INTERVENTIONS:
Behavioral: Mindful Moms — Twelve 75 minutes weekly group sessions involving gentle yoga practices designed for pregnant women, led by experienced yoga teachers.
  Arms: Mindful Moms
Behavioral: Prenatal Education — Twelve 75 minutes weekly group sessions involving prenatal education (for example, what to expect during your pregnancy, during labor and delivery, and after the delivery of your child).
  Arms: Prenatal Education

SUMMARY:
The purpose of this study is to test whether a program called "Mindful Moms" can be helpful for specific measures of mood and health in pregnant women with depressive symptoms, compared to group-based education workshops.

DETAILED DESCRIPTION:
The Mindful Moms Study is a randomized controlled trial, in which participants will be randomly assigned (like the flip of a coin) to either the "Mindful Moms" group (12 weeks of group-based prenatal yoga) or the "Prenatal Education Circle" group (12 weeks of group-based prenatal education). 200 pregnant women will participate over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant woman at 12-26 weeks gestation at baseline visit;
2. defined as minority (e.g., Black/ African American, Hispanic/ Latino, Native American, etc) and/or annual household income at qualification level for Women, Infants, & Children [WIC] benefits in Virginia and/or educational attainment ≤high school education;
3. ≥age 18;
4. current depressive symptoms, as defined by a score ≥7 on the Edinburgh Postnatal Depression Scale (EPDS);
5. able to read, write, and understand English;
6. has not been told by a healthcare provider to avoid physical activity;
7. has not engaged in a consistent (once/week or more) yoga-based practice during the current pregnancy.

Exclusion Criteria: Does not meet the inclusion criteria above.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 200 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive symptom severity | Baseline to postpartum, about 8 months
  Depressive symptoms will be assessed using the Edinburgh Postnatal Depression Scale (EPDS). The EDPS is a widely used and validated measure of depressive symptoms, with 10 questions appropriate for the prenatal and postpartum woman; a score ≥10 (range 0-30) suggests possible depressive symptoms.

SECONDARY OUTCOMES:
Change in anxiety | Baseline to postpartum, about 8 months
  Anxiety will be assessed using the Perinatal Anxiety Screening Scale (PASS); scores range from 0-93, high scores indicate higher levels of anxiety.
Change in stress | Baseline to postpartum, about 8 months
  Stress will be assessed using the JHP Contextualized Stress Measure. The JHP measures the stressors and coping mechanisms to which women are exposed to, with a range of score from 25-125 (higher score indicates higher stress)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kinser, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kinser PA, Bodnar-Deren S, Amstadter AB, Lapato DM, Thacker LR, Johnson JA, Aubry C, Johnson A, Gault C, Hill-Thomas A, Russell S, Lanni S, Freeman A. Study protocol for the Mindful Moms Study: A randomized controlled trial evaluating a mindful movement intervention for marginalized pregnant people experiencing depression. Contemp Clin Trials. 2023 Sep;132:107302. doi: 10.1016/j.cct.2023.107302. Epub 2023 Jul 25. PMID 37500008